CLINICAL TRIAL: NCT03661437
Title: Light Therapy to Prevent Frailty in Older Men With Prostate Cancer on Hormonal Therapy: A Pilot RCT
Brief Title: Systemic Light Exposure in Preventing Frailty in Older Patients With Prostate Cancer on Hormonal Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18140; NCI-2018-01868 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18140 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (BWL) (Experimental): Patients wear an Actiwatch for 5 days at baseline, 3 months and 6 months. Beginning 1-4 weeks after first anti-androgen therapy, patients undergo BWL treatment using Luminette glasses for 30 minutes every morning for 3-6 months.
  Interventions: Device: Actigraph; Other: Questionnaire Administration; Procedure: Systematic Light Exposure
- Arm II (DWL) (Experimental): Patients wear an Actiwatch for 5 days at baseline, 3 months and 6 months. Beginning 1-4 weeks after first anti-androgen therapy, patients undergo DWL treatment using Luminette glasses for 30 minutes every morning for 3-6 months.
  Interventions: Device: Actigraph; Other: Questionnaire Administration; Procedure: Systematic Light Exposure

INTERVENTIONS:
Device: Actigraph — Wear Actiwatch
  Other Names: Actigram
Other: Questionnaire Administration — Ancillary studies
Procedure: Systematic Light Exposure — Undergo BWL treatment
  Other Names: sLE
  Arms: Arm I (BWL)
Procedure: Systematic Light Exposure — Receive DWL treatment
  Other Names: sLE
  Arms: Arm II (DWL)

SUMMARY:
This pilot trial studies how well systemic light exposure works in preventing frailty in older patients with prostate cancer on hormonal therapy. Hormone therapy causes many symptoms of frailty in older men including fatigue, slower time to walk a specified distance, reduced activity levels, loss of lean muscle, and muscle weakness. It is not yet known if systemic light exposure may reduce frailty in older prostate cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if bright white light (BWL), compared to dim white light (DWL), significantly prevents frailty development in older prostate cancer (PC) patients following prostate anti-androgen therapy initiation.

II. Determine if BWL, compared to DWL, significantly increases functional performance and physical activity levels, yields significant reductions in fatigue, lowers body mass index (BMI), and reduces weakness in older PC patients following prostate anti-androgen therapy initiation.

EXPLORATORY OBJECTIVE:

I. Examine the feasibility of collecting and storing clinically-usable bio-measures for future analysis in patients at baseline and if available at 6 months, including blood samples (inflammatory markers), and salivary swabs (genetics, genomics, cortisol circadian rhythms).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (BWL): Patients wear an Actiwatch for 5 days at baseline, 3 months and 6 months. Beginning 1-4 weeks after first anti-androgen therapy, patients undergo BWL treatment using Luminette glasses for 30 minutes every morning for 3-6 months.

ARM II (DWL): Patients wear an Actiwatch for 5 days at baseline, 3 months and 6 months. Beginning 1-4 weeks after first anti-androgen therapy, patients undergo DWL treatment using Luminette glasses for 30 minutes every morning for 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer (PC) patients who are starting androgen deprivation therapy (ADT), abiraterone, or enzalutamide with plans to continue for at least six months with minimal evidence of disease burden in accordance with current standards of care.
* A life expectancy of 6 months or longer.
* All subjects must have the ability to understand and the willingness to sign a written or electronic informed consent.

Exclusion Criteria:

* Significant pre-existing frailty precluding completion of baseline assessments.
* Other active malignancies
* Previous use of radiation therapy within the year prior to consent.
* Widely metastatic disease.
* Confounding serious medical illnesses which causes frailty.
* Severe sleep disorders.
* Eye diseases which limit the ability of light to be processed.
* Severe psychological impairment.
* Current employment in night shift work.
* Previous use of light therapy to alleviate fatigue or depressive symptoms.
* Secondary cancer diagnosis within the past 5 years.
* Plans to travel across meridians during treatment.
* Uncontrolled illness including ongoing or active infection in disease status patients.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Physical performance in older prostate cancer (PC) patients following prostate anti-androgen therapies initiation | Up to 6 months
  Will be assessed using Short Physical Performance Battery (SPPB). Will be evaluated using a repeated measures mixed linear model.
Frailty development in older PC patients following prostate anti-androgen therapies initiation | Up to 6 months
  Will be assessed using SPPB. Will be evaluated using a repeated measures mixed linear model.

SECONDARY OUTCOMES:
Fatigue level | Up to 6 months
  Will be measured using the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue. Will be evaluated using a repeated measures mixed linear model.
Physical performance | Up to 6 months
  Will be assessed by measuring the waist and hip circumference using a fabric measuring tape to determine the circumference of the waist (centered at the umbilicus) and hip (centered on the greater trochanter). Will be evaluated using a repeated measures mixed linear model.
Hand-grip strength measured using hand-held dynamometer | Up to 6 months
  Muscle weakness will be measured by grip strength. Will be evaluated using a repeated measures mixed linear model.
Instrumental activities of daily living (IADL) scale | Up to 6 months
  Will be evaluated using a repeated measures mixed linear model.
Activity level | Up to 6 months
  Activity counts will be recorded with the Actiwatch Spectrum Plus for five days at each time-point. Will be evaluated using a repeated measures mixed linear model.

OTHER OUTCOMES:
Collecting and storing clinically-usable bio-measures | Baseline up to 6 months
  Blood samples and saliva swaps will be collected for future analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William Dale, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States